CLINICAL TRIAL: NCT02129153
Title: Linking Families Together Study- A Randomized Trial to Raise Parental Monitoring
Acronym: LIFT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Dr. Mitchell Wong, Associate Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: IRB#13-001638
Record Dates: First submitted 2014-04-30; First posted 2014-05-02 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Adolescent Behaviors; Substance Abuse
Keywords: Randomized controlled trial; Population, School Age
MeSH Terms: conditions — Adolescent Behavior; Substance-Related Disorders | interventions — Lifting

STUDY DESIGN:
Who Masked: Participant
Masking Description: Participants in the study do not know if they are in the intervention group.
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LIFT (Parent information) (Experimental): LIFT (Parent information): during their child's 7th and 8th grade years research staff will 1. communicate with parents about their child's academic and behavioral performance in school, roughly twice-monthly 2. invite parents to participate in a 2-hour parent support session to help teach parents to communicate better with their child and support better academic and behavioral performance in school
  * students take a baseline survey then 3 surveys (one/year)
  * parents take a baseline survey then 2 surveys (one/year)
  Interventions: Behavioral: LIFT (Parent Information)
- Usual care group (No Intervention): Usual care control group/No Intervention consists of neither communication of academic information to parents nor invitation to parent support sessions.
  * students take a baseline survey then 3 surveys (one/year)
  * parents take a baseline survey then 2 surveys (one/year)

INTERVENTIONS:
Behavioral: LIFT (Parent Information) — 1. Parents will receive specific information about class assignments that the student missed or about poor performance on tests/quizzes. Parents will also be notified about behavioral problems, such as poor attention and class disruption. RA will communicate with parents in Spanish or English by text message, phone, email according to the parents preference for communication
  2. Parents will be invited to parenting seminars to discuss parenting strategies regarding what to do with their child's academic and behavioral information once they receive it from research staff. Sessions will take place at school and last 2 hours. Multiple sessions will be offered throughout the academic year and parents may attend as many sessions as they wish.
  Other Names: Information/ Linking Families Together (LIFT)
  Arms: LIFT (Parent information)

SUMMARY:
In this study, we will evaluate the efficacy and sustainability of the Linking Families Together (LIFT) intervention to improve parental monitoring during the transition from middle to high school a particularly risky time for students' academic performance and health behaviors. This study is based in middle schools around Los Angeles County a region with a high prevalence of teen risky health behaviors.

The aims of our study are:

1. To conduct a randomized trial of the LIFT intervention and examine whether providing detailed academic information to parents during their child's 7th and 8th grade increases parental monitoring at the end of the two year intervention and one year follow up. We will partner with 3-10 middle schools and recruit 500 student-parent dyads: 250 will be randomized to the intervention arm and 250 to the usual care control group.
2. To determine whether the LIFT intervention improves students' academic outcomes, as measured by grades, attendance, and standardized test scores at the end of the two year intervention and one year follow up.
3. To evaluate whether the LIFT intervention lowers rates of adolescent risky health behaviors, specifically substance use (alcohol, marijuana, inhalants, and other drugs) at the end of the two year intervention and one year follow up.

DETAILED DESCRIPTION:
Despite parental monitoring and school involvement being among the most important protective factors leading to positive teen academic and health trajectories, few theoretically based rigorously evaluated interventions test strategies to support low income parents as their adolescents transition from middle to high school, a particularly risky time for students' academic and health behaviors.

In a successful pilot study, student's missing assignments information was communicated directly to parents. Intervention parents were nearly twice as likely to report their child not telling them enough about his or her school work than control parents. After just 6 months, intervention students had a 0.19 standard deviation increase in GPA over the control group and 0.20 standard deviation higher standardized math test score.

In the proposed study, we will evaluate the efficacy and sustainability of an intervention to improve parental monitoring and thus improve academic outcomes and reduce risky health behaviors. The adapted intervention will also include sessions for parents to build positive parent-child communication and awareness of school expectations.

We propose a randomized controlled trial with 2 arms examining whether providing parents detailed information on their child's academic and behavioral performance in school in combination with basic parenting support, increases parental monitoring for low-income, minority families. We hypothesize that better parental monitoring will lead to improved academic and behavioral performance. Using this design we can determine whether the impact of the information and parenting intervention is also protective of teens engaging in risky health behaviors. We will compare the experimental and control group parents to examine whether providing high-quality academic information to parents of middle school students increases parental monitoring, student academic performance, and teen health outcomes during middle school and beyond.

If the intervention boosts adolescent academic and health outcomes as hypothesized, the results of the proposed study offer schools low-cost strategies to simultaneously positively influence student academic and health trajectories. These findings have the potential to stimulate new research to improve health through innovative interventions to bolster parent teen relationships for gains accrued throughout the life span.

The aims of our study are:

1. To conduct a randomized trial of the LIFT intervention and examine whether providing detailed academic information to parents during their child's 7th and 8th grade increases parental monitoring at the end of the two year intervention and one year follow up. We will partner with 3-10 middle schools and recruit 500 student-parent dyads: 250 will be randomized to the intervention arm and 250 to the usual care control group.
2. To determine whether the LIFT intervention improves students' academic outcomes, as measured by grades, attendance, and standardized test scores at the end of the two year intervention and one year follow up.
3. To evaluate whether the LIFT intervention lowers rates of adolescent risky health behaviors, specifically substance use (alcohol, marijuana, inhalants, and other drugs) at the end of the two year intervention and one year follow up.

Thus the proposed study builds on and extends the earlier pilot study by recruiting more middle schools around Los Angeles, offering parents additional supports through parenting workshops, and assessing the program's impact on adolescent behavioral outcomes. Successfully implementing this study will allow us to demonstrate feasibility for a future randomized controlled trial and assess effect size for parental monitoring and health outcomes.

ELIGIBILITY:
Inclusion Criteria:

* For adults, must be a parent/guardian of a student at a participating middle school
* For minors, must be a student at a participating middle school
* Must speak English or Spanish
* Entering 7th grade in Fall 2014 at one of the middle schools participating in the study

Exclusion Criteria:

* None

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 318 (Actual)
Dates: Start 2014-09-01; Primary Completion 2016-06-30 (Actual); Study Completion 2016-08-01 (Actual)

PRIMARY OUTCOMES:
Change from baseline in student 30 day alcohol use | baseline, two year, three year (i.e. one year follow up)
  Student self report: During the past 30 days, on how many days did you have at least one drink of alcohol?

SECONDARY OUTCOMES:
Change from baseline in student 30 day marijuana use | baseline, two year, three year (i.e. one year follow up)
  Student self report: During the past 30 days, on how many days did you use marijuana?
Change from baseline in parental monitoring | baseline, two year, three year (i.e. one year follow up)
  Student completing validated 9-item parental monitoring scale
Change from baseline in student standardized test scores | baseline, two year, three year (i.e. one year follow up)
  Student standardized test scores

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell D Wong, MD PhD, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bergman P, Dudovitz RN, Dosanjh KK, Wong MD. Engaging Parents to Prevent Adolescent Substance Use: A Randomized Controlled Trial. Am J Public Health. 2019 Oct;109(10):1455-1461. doi: 10.2105/AJPH.2019.305240. Epub 2019 Aug 15. PMID 31415193